CLINICAL TRIAL: NCT00962390
Title: Randomized, Double Blind, Multicenter, Placebo Controlled, Proof of Concept Trial to Assess the Efficacy and Safety of 4 Weeks Treatment With AUS 131 (S Equol) on Benign Prostatic Hyperplasia
Brief Title: Efficacy and Safety of S-Equol on Men With Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ausio Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUS CT04
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Equol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 150mg S-equol (Experimental)
  Interventions: Drug: S-equol
- 50mg S-equol (Experimental)
  Interventions: Drug: S-equol
- 10 mg S-equol (Experimental)
  Interventions: Drug: S-equol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-equol — 10mg S-equol 50mg S-equol, & 150mg S-equol
  Other Names: AUS-131
  Arms: 10 mg S-equol; 150mg S-equol; 50mg S-equol
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of S-equol in men with benign prostatic hyperplasia.

DETAILED DESCRIPTION:
The study is a phase 2a, randomized, double blind, multicenter, placebo controlled, parallel group, proof of concept study comparing the efficacy, safety, and acceptability of S-equol to placebo in patients with benign prostatic hyperplasia. The study objective is to examine a dose response of 3 dose levels of S equol versus placebo on prostate specific antigen concentrations in patients with benign prostatic hyperplasia. The safety of S-equol will be evaluated during the study.

ELIGIBILITY:
Inclusion Criteria:

* Is male > 50 years of age at Screening.
* Has a normal digital rectal exam with the exception of prostate enlargement.
* Has suffered from symptoms of BPH for at least the 6 months before Screening.
* Has a prostate volume ≥ 20 mL and ≤ 70 mL as assessed by ultrasound.
* Has a serum PSA concentration > 1.5 ng/mL and ≤ 10 ng/mL at Screening.
* Has an IPSS > 13 at Screening and Baseline.
* Has a Qmax > 5 cc/sec and < 15 cc/sec with a voided volume ≥ 125 cc at Screening (and Baseline, if applicable).

Exclusion Criteria:

* Has a known history of allergic reaction or clinically significant intolerance to ingredients of the study drug.
* Neurogenic bladder dysfunction.
* Has bladder neck contracture or urethral stricture.
* Has acute or chronic prostatitis or urinary tract infection.
* Has, or has a history of, prostate cancer or carcinoma of the prostate suspected on digital rectal exam or transrectal ultrasound, or has a serum PSA concentration > 10 ng/mL; patients with a PSA concentration > 4 ng/mL and ≤ 10 ng/mL must have prostate cancer ruled out to the satisfaction of the investigator.
* Has a residual void volume > 250 mL.
* Has any clinically significant unstable condition that, in the opinion of the investigator, could compromise the patient's welfare, ability to communicate with the study staff, or otherwise contraindicate study participation.
* Shows presence of any manifest premalignant or malignant disease except treated skin cancers (except melanoma).
* Has a history of smoking more than 5 cigarettes daily within the year before Screening.
* Has resting systolic blood pressure (BP) > 160 mmHg or < 90 mmHg, or diastolic BP > 90 mmHg or < 60 mmHg at Screening.
* Has bladder stones as detected by ultrasound.
* Has hematuria of unknown etiology.
* Had previous prostate surgery or other invasive treatment for BPH.
* Had prior radiation to the pelvis.
* Has Parkinson's disease or multiple sclerosis.
* Had stroke or myocardial infarction within 5 months before Baseline.
* Has abnormal screening electrocardiogram (ECG) or unstable angina or severe congestive heart failure.
* Has active liver disease renal insufficiency with creatinine > 1.7 mg/dL, or clinically significant abnormal hemoglobin, white blood cell count, or platelet count.
* Has a history of postural hypotension or has a fall in systolic BP > 20 mm Hg after 2 minutes in a standing position.
* Received alpha blocker therapy within 28 days before Baseline.
* Received androgens, anti androgens, 5 alpha reductase inhibitors, or luteinizing hormone releasing hormone (LHRH) analogs within 3 months before Baseline.
* Received tricyclic antidepressants or plant extracts (e.g., saw palmetto) within 1 month before Baseline.
* Received sedating antihistamines, sympathomimetics, or anticholinergics within 1 week before Baseline.
* Has initiated new use (i.e., within the past 4 weeks before Screening) or otherwise are not on stable doses of phosphodiesterase 5 inhibitors during the 4 weeks before Screening.
* Has known or suspected history of alcoholism or drug abuse or misuse within the last 5 years.
* Is considered by the investigator, for any reason (including, but not limited to, the risks described as precautions, warnings, and contraindications in the current version of the Clinical Investigator's Brochure for AUS 131 [S equol]), to be an unsuitable candidate to receive the study drug.
* Has tested positive on the urine drug screen.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Bergner, MD, Principal Investigator — Tampa Bay Medical Research
Locations (15):
- United States (5):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - South Florida Medical Research, Aventura, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Advanced Clinical Research, West Jordon, Utah
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
- India (10):
  - Samved Hospital, Ahmedabad
  - M S Ramaiah Memorial Hospital, Bangalore
  - St. John's Medical College Hospital, Bangalore
  - G S Medical College and KEM Hospital, Delhi
  - Indraprastha Apollo Hospital, Delhi
  - V M Medical College and Safdarjung Hospital, Delhi
  - SMS Hospital, Jaipur
  - A J Hospital and Research Center, Mangalore
  - Inamdar Multispecialty Hospital, Pune
  - Ruby Hall Clinic, Pune

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 4 centers in Australia, 10 centers in India, and 8 centers in the United States from February 2010 to August 2015. The first participant was enrolled in August 2010, and the last participant was enrolled in August 2015.
Groups:
- S-equol 10 mg BID: Experimental: S-equol
  Participants received S-equol 10 mg capsule orally twice daily (20 mg total daily dose) for 4 weeks.
- S-equol 50 mg BID: Experimental: S-equol
  Participants received S-equol 50 mg capsule orally twice daily (100 mg total daily dose) for 4 weeks.
- S-equol 150 mg BID: Experimental: S-equol
  Participants received S-equol 150 mg capsule orally twice daily (300 mg total daily dose) for 4 weeks.
- Placebo BID: Placebo Comparator: Placebo
  Participants received S-equol placebo capsule matching S-equol orally twice daily for 4 weeks.
Period: Overall Study
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Started | 29 | 29 | 29 | 29
Completed | 25 | 26 | 25 | 28
Not Completed | 4 | 3 | 4 | 1
Not completed — Adverse Event | 0 | 0 | 3 | 1
Not completed — Lost to Follow-up | 2 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who took at least one (1) dose of investigational product were included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID | Total
Number analyzed (Participants) | 28 | 29 | 29 | 29 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (9.1) | 64.6 (6.5) | 63.1 (8.8) | 62.7 (7.7) | 63.4 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 28 | 29 | 29 | 29 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 3 | 8
  Not Hispanic or Latino | 26 | 28 | 27 | 26 | 107
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 10 | 11 | 11 | 13 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 0 | 9
  White | 14 | 15 | 15 | 16 | 60
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Prostate specific antigen (PSA) concentration [Mean (Standard Deviation); unit: ng/mL] — Population: Participants who had taken at least one (1) dose of investigational product and had a baseline value of interest.
  ng/mL
    number analyzed (Participants) | 28 | 28 | 28 | 29 | 113
    (all) | 3.509 (2.241) | 3.308 (1.796) | 3.210 (1.075) | 3.514 (1.860) | 3.386 (1.775)
Prostate Volume [Mean (Standard Deviation); unit: mL] — Population: Participants who had taken at least one (1) dose of investigational product and had a baseline value of interest.
  mL
    number analyzed (Participants) | 28 | 28 | 28 | 29 | 113
    (all) | 43.46 (13.47) | 44.79 (14.27) | 40.83 (11.40) | 41.41 (11.39) | 42.61 (12.62)
Post Void Residual Urine Volume [Mean (Standard Deviation); unit: mL] — Population: Participants who had taken at least one (1) dose of investigational product and had a baseline value of interest.
  mL
    number analyzed (Participants) | 28 | 28 | 28 | 29 | 113
    (all) | 74.59 (60.45) | 62.00 (55.93) | 61.38 (60.37) | 89.07 (56.01) | 71.91 (58.55)
Qmax Result [Mean (Standard Deviation); unit: mL/second] — Population: Participants who had taken at least one (1) dose of investigational product and had a baseline value of interest.
  mL/second
    number analyzed (Participants) | 28 | 28 | 28 | 29 | 113
    (all) | 10.22 (3.13) | 10.27 (3.29) | 11.17 (3.30) | 10.98 (3.59) | 10.66 (3.32)
Void Volume [Mean (Standard Deviation); unit: mL] — Population: Participants who had taken at least one (1) dose of investigational product and had a baseline value of interest.
  mL
    number analyzed (Participants) | 28 | 28 | 28 | 29 | 113
    (all) | 229.21 (128.59) | 245.75 (111.49) | 243.54 (115.54) | 261.48 (86.07) | 245.14 (110.39)
Dihydrotestosterone [Mean (Standard Deviation); unit: pg/mL] — Population: Participants who had taken at least one (1) dose of investigational product and had a baseline value of interest.
  pg/mL
    number analyzed (Participants) | 28 | 28 | 26 | 27 | 109
    (all) | 496.2 (425.2) | 533.6 (388.5) | 534.7 (467.4) | 446.1 (185.5) | 502.6 (378.3)
Luteinizing Hormone [Mean (Standard Deviation); unit: IU/L] — Population: Participants who had taken at least one (1) dose of investigational product and had a baseline value of interest.
  IU/L
    number analyzed (Participants) | 28 | 28 | 26 | 28 | 110
    (all) | 5.4 (4.2) | 5.1 (2.5) | 6.5 (4.1) | 5.9 (2.8) | 5.7 (3.5)
Testosterone, Total [Mean (Standard Deviation); unit: nmol/L] — Population: Participants who had taken at least one (1) dose of investigational product and had a baseline value of interest.
  nmol/L
    number analyzed (Participants) | 28 | 28 | 26 | 28 | 110
    (all) | 442.6 (311.7) | 319.9 (248.0) | 340.6 (180.9) | 372.7 (202.0) | 369.5 (243.2)
Total International Prostate Symptom Score (I-PSS) [Mean (Standard Deviation); unit: units on a scale] — The I-PSS is based on the answers to 7 questions concerning urinary symptoms and one question concerning the quality of life. Each question concerning urinary symptoms allows the subject to choose 1 out of 6 answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can, therefore, range from 0 (asymptomatic) to 35 (very symptomatic). Population: Participants who had taken at least one (1) dose of investigational product and had a baseline value of interest.
  units on a scale
    number analyzed (Participants) | 28 | 28 | 28 | 28 | 112
    (all) | 21.11 (5.24) | 23.64 (4.57) | 21.50 (4.59) | 21.32 (5.21) | 21.89 (4.96)
Total Danish Prostatic Symptom Score (DAN-PSS-1) [Mean (Standard Deviation); unit: units on a scale] — The DAN-PSS-1 is a self-administered quality-of-life questionnaire comprising 12 questions related to lower urinary tract symptoms (bladder storage and voiding function), and 3 questions related to sexual function (symptom score). All answers for symptom and bothersomeness were classified in a 4-ranked scale from 0 (absence of symptoms or no impact on daily life) to 3 (the maximum severity of symptoms or impact on daily life). A weighted score was then calculated to give a total score that ranged from 0 to 108, where higher scores represented worsening symptoms and bothersomeness. Population: Participants who had taken at least one (1) dose of investigational product and had a baseline value of interest.
  units on a scale
    number analyzed (Participants) | 28 | 28 | 29 | 29 | 114
    (all) | 26.1 (10.9) | 33.5 (15.3) | 27.2 (15.5) | 31.1 (19.1) | 29.5 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 4 in Prostate Specific Antigen (PSA) Concentration.
Description: Prostate specific antigen is considered to be the most sensitive measure of S-equol effects on the prostate, due to the expected effects of S-equol on the androgen receptor axis. In this proof-of-concept study, a population of 124 male subjects was estimated to achieve approximately 104 completed subjects (based on an estimated drop-out rate of 15%) to examine the dose-response compared to placebo. A sample size of 26 subjects in each treatment arm was considered to be adequate to observe a trend in this proof-of-concept study.
Time Frame: 4 weeks
Population: All Participants who received at least 1 dose of study drug and who had a post-dose PSA assessment at Week 4.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 25 | 26 | 24 | 29
ng/mL | -0.1 (0.3) | -0.1 (0.3) | -0.3 (0.3) | -0.4 (0.3)
Statistical Analysis 1: Comparison: S-equol 10 mg BID vs Placebo BID; Week 4, Treatment Effect; Test type: Superiority or Other; p = 0.4678, ANCOVA — Statistical testing was 2-sided and the 5% significant level was used; The ANCOVA included Baseline as covariate and factors for treatment and site; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.5 to 1.1] — S-equol treatment group minus placebo group
Statistical Analysis 2: Comparison: S-equol 50 mg BID vs Placebo BID; Week 4, Treatment Effect; Test type: Superiority or Other; p = 0.4892, ANCOVA — Statistical testing was 2-sided and the 5% significant level was used; The ANCOVA included Baseline as covariate and factors for treatment and site; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.5 to 1.1] — S-equol treatment group minus placebo group
Statistical Analysis 3: Comparison: S-equol 150 mg BID vs Placebo BID; Week 4, Treatment Effect; Test type: Superiority or Other; p = 0.8185, ANCOVA — Statistical testing was 2-sided and the 5% significant level was used; The ANCOVA included Baseline as covariate and factors for treatment and site; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.8 to 1.0] — S-equol treatment group minus placebo group

2. Secondary Outcome: Change in Prostate Volume From Baseline at Week 4
Description: Prostate size as measured by prostate volume as assessed by transrectal ultrasound.
Time Frame: 4 weeks
Population: All randomized subjects who received at least 1 dose of investigational product starting at Baseline, and who had at least 1 post-dose assessment of interest.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 24 | 26 | 22 | 28
mL
  Week 4 Values | 40.03 (12.10) | 45.53 (15.36) | 39.16 (10.67) | 39.73 (13.98)
  Change from Baseline | -3.03 (5.28) | -0.25 (8.29) | -1.72 (7.31) | -1.74 (5.10)

3. Secondary Outcome: Change in Qmax From Baseline at Week 4
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 25 | 26 | 23 | 28
mL/sec
  Week 4 Values | 11.00 (5.87) | 10.10 (5.41) | 14.40 (5.70) | 13.40 (6.57)
  Change from Baseline | 0.96 (4.74) | -0.09 (6.13) | 2.49 (6.25) | 2.25 (6.63)

4. Secondary Outcome: Categorical Change in Qmax From Baseline at Week 4
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 25 | 26 | 23 | 28
Participants
  Week 4 Values, <=2 mL/sec | 17 | 19 | 13 | 17
  Week 4 Values, >2 mL/sec | 8 | 7 | 10 | 11

5. Secondary Outcome: Percent Change in Qmax From Baseline at Week 4
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 25 | 26 | 22 | 28
Participants
  Week 4 Values, <=30% | 18 | 22 | 13 | 19
  Week 4 Values, >30% | 7 | 4 | 9 | 9

6. Secondary Outcome: Change in Void Volume From Baseline at Week 4
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 25 | 26 | 22 | 28
mL
  Week 4 Values | 235.04 (124.23) | 191.50 (88.79) | 312.09 (187.12) | 266.32 (119.92)
  Change from Baseline | 4.04 (128.97) | -58.00 (116.23) | 72.18 (154.08) | 7.46 (134.59)

7. Secondary Outcome: Change in Post-Void Residual Volume From Baseline at Week 4
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 25 | 26 | 23 | 28
mL
  Week 4 Values | 77.90 (96.73) | 83.54 (96.98) | 52.46 (68.14) | 85.90 (81.25)
  Change from Baseline | 2.51 (93.12) | 17.08 (93.73) | -18.22 (69.97) | -6.28 (73.29)

8. Secondary Outcome: Change in in Dihydrotestosterone Concentration From Baseline at Week 4
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 22 | 24 | 22 | 27
pg/mL
  Week 4 Values | 584.7 (567.0) | 532.4 (483.1) | 616.6 (661.9) | 502.4 (434.5)
  Change from Baseline: number analyzed (Participants) | 22 | 23 | 20 | 25
  Change from Baseline | 64.2 (313.1) | -6.2 (139.9) | 68.1 (488.9) | -14.5 (72.9)

9. Secondary Outcome: Change in Luteinizing Hormone Concentration From Baseline at Week 4
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 23 | 26 | 23 | 28
IU/L
  Week 4 Values | 4.4 (2.6) | 6.0 (3.4) | 6.1 (4.1) | 5.9 (2.9)
  Change from Baseline: number analyzed (Participants) | 23 | 25 | 21 | 27
  Change from Baseline | -0.6 (2.2) | 1.1 (2.5) | -0.3 (2.4) | 0.0 (2.0)

10. Secondary Outcome: Change in Total Testosterone Concentration From Baseline at Week 4
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 23 | 26 | 23 | 28
nmol/L
  Week 4 Values | 449.9 (283.7) | 310.3 (204.2) | 314.0 (177.2) | 351.3 (176.8)
  Change from Baseline: number analyzed (Participants) | 23 | 25 | 21 | 27
  Change from Baseline | -8.1 (116.4) | -2.6 (173.8) | 3.7 (93.9) | -34.4 (128.4)

11. Secondary Outcome: Participants Assessment of Nocturia at Week 4
Description: Participants were asked to rate their change in nocturia (number of times you wake from sleep to urinate) since the Baseline Visit.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: number of times to urinate at night
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 27 | 28 | 26 | 29
number of times to urinate at night | 3.0 [1 to 6] | 3.0 [1 to 5] | 3.0 [2 to 7] | 3.0 [1 to 4]

12. Secondary Outcome: Investigators Assessment of Nocturia at Week 4
Description: Investigators were asked to rate participant's change in nocturia since the Baseline Visit.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: number of times urinated at night
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 25 | 26 | 24 | 28
number of times urinated at night | 3.0 [1 to 6] | 3.0 [1 to 5] | 3.0 [1 to 4] | 3.0 [1 to 4]

13. Secondary Outcome: Change in I-PSS Total Score From Baseline at Week 4
Description: The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of 6 answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic). The first seven questions of the I-PSS are identical to the questions appearing on the American Urological Association (AUA) Symptom Index which currently categorizes symptoms as follows: Mild (symptom score less than of equal to 7); Moderate (symptom score range 8-19); and Severe (symptom score range 20-35). A reduction in I-PSS Total Score is consistent with improvement in symptoms of BPH.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 27 | 28 | 26 | 29
units on a scale
  Week 4 Values | 15.56 (5.35) | 17.46 (5.79) | 17.54 (6.96) | 15.07 (7.62)
  Change from Baseline: number analyzed (Participants) | 27 | 28 | 26 | 28
  Change from Baseline | -5.81 (7.56) | -6.18 (5.55) | -4.15 (6.42) | -5.96 (5.83)

14. Secondary Outcome: Change in DAN Prostate Symptom Scale From Baseline at Week 4
Description: The questionnaire is made up of two kinds of questions: intensity of a symptom and bothersomeness of a symptom. Prostate symptoms are addressed in questions 1 - 12 and sexual function in questions 13 - 15. Patients indicate how intense/frequent (scoring 0, 1, 2, or 3; where 0 represents the best case and 3 the worst case) and how bothersome the symptom (scoring 0, 1, 2, or 3; where 0 is 'not at all' and 3 is 'very much'). DAN-PSS total and DAN-PSS total sexual function score were calculated by multiplying the frequency score by the trouble score of each symptom, and then adding the resulting figures. The possible values of DAN-PSS total ranged from 0 to 108 and of DAN-PSS total sexual function score ranged from 0 to 27. A reduction in DAN-PSS total and/or sexual function score is consistent with improved BPH symptoms/sexual functioning.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
Number analyzed (Participants) | 27 | 28 | 27 | 27
units on a scale
  Total Score, Week 4 Values | 17.7 (10.9) | 22.1 (14.9) | 22.7 (14.6) | 20.3 (20.8)
  Total Score, Change from Baseline | -8.2 (12.9) | -11.5 (15.4) | -4.7 (12.0) | -10.0 (15.2)
  Sexual Function Score, Week 4 Values: number analyzed (Participants) | 19 | 19 | 20 | 20
  Sexual Function Score, Week 4 Values | 2.2 (3.1) | 4.2 (5.4) | 5.6 (3.8) | 4.7 (5.9)
  Sexual Function Score, Change from Baseline: number analyzed (Participants) | 17 | 17 | 19 | 18
  Sexual Function Score, Change from Baseline | -0.3 (1.6) | 0.2 (2.9) | -1.2 (4.7) | 0.3 (2.5)

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of signing of the ICF through the Follow-up Visit (Visit 6) or Early Termination Visit (whichever occurred first), up to Day 56±2 days.
Description: The investigator monitored and/or asked about or evaluated adverse events (AEs) using non-leading questions at each visit or evaluation. The occurrence of all AEs were documented in the Adverse Event Case Report Form.
Groups:
- S-equol 10 mg BID: Experimental: S-equol
  Participants received S-equol 10 mg capsule orally twice daily (20 mg total daily dose) for 4 weeks.
  At-risk Participants were subjects who received at least one dose of S-at any time during the study.
- S-equol 50 mg BID: Experimental: S-equol
  Participants received S-equol 50 mg capsule orally twice daily (100 mg total daily dose) for 4 weeks.
  At-risk Participants were subjects who received at least one dose of S-at any time during the study.
- S-equol 150 mg BID: Experimental: S-equol
  Participants received S-equol 150 mg capsule orally twice daily (300 mg total daily dose) for 4 weeks.
  At-risk Participants were subjects who received at least one dose of S-at any time during the study.
- Placebo BID: Placebo Comparator: Placebo
  Participants received S-equol placebo capsule matching S-equol orally twice daily for 4 weeks.
  At-risk Participants were subjects who received at least one dose of S-at any time during the study.
Arm/Group | S-equol 10 mg BID | S-equol 50 mg BID | S-equol 150 mg BID | Placebo BID
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/29 | 1/29 | 0/29
Other Adverse Events (participants affected / at risk) | 6/28 | 5/29 | 8/29 | 5/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | S-equol 10 mg BID (N=28) | S-equol 50 mg BID (N=29) | S-equol 150 mg BID (N=29) | Placebo BID (N=29)
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | S-equol 10 mg BID (N=28) | S-equol 50 mg BID (N=29) | S-equol 150 mg BID (N=29) | Placebo BID (N=29)
Vision Blurred (Eye disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 1 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Paraesthesia of genital male (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less